CLINICAL TRIAL: NCT02714738
Title: The Ultrasound Guided Infraclavicular Block: Decreased Incidence of Tourniquet Pain, Compared to Axillary Brachial Plexus Block?
Brief Title: Infraclavicular Block: Decreased Incidence of Tourniquet Pain, Compared to Axillary Brachial Plexus Block?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cork University Hospital (Other)
Responsible Party: Principal Investigator, Dr. David Brenner, Principial Investigator, Cork University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TP-ICB-ABPB
Record Dates: First submitted 2016-03-16; First posted 2016-03-21 (Estimated); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Tourniquet Pain
Keywords: Brachial plexus block; Regional anesthesia; Ultrasound

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Infraclavicular Block (Experimental): The patient will be positioned supine. The operating limb may be positioned abducted or adducted by side depending on operator preference and patient factors. After standard preparation, the needle will be directed towards the target area using an in-plane, short-axis technique. Local anaesthetic (lidocaine 2% with epinephrine 1:200.000) will be injected posterior to the artery with the intention achieving the U shape, cranio-postero-caudal spread. Local anaesthetic will be deposited to the lateral and medial cords as well, if required. The total dose of the local anaesthetic will be 20-30 ml, as clinically indicated.
  Interventions: Procedure: Ultrasound guided peripheral nerve block
- Axillary Brachial Plexus Block (Experimental): The patient will be positioned supine with the operative upper limb extended, flexed at the elbow, rested on a pillow to expose the axilla. After standard preparation, the needle will be directed towards the target area using an in-plane, short-axis technique. All four nerves in the axillary region are being blocked. The local anesthetic (lidocaine 2% with epinephrine 1:200.000, 15-25 ml) will be divided among the four nerves as clinically indicated by the spread, but at least 3 ml applied to each nerve.
  Interventions: Procedure: Ultrasound guided peripheral nerve block

INTERVENTIONS:
Procedure: Ultrasound guided peripheral nerve block — Ultrasound guided peripheral nerve block

SUMMARY:
The purpose of this study is to determine whether the incidence of tourniquet pain is decreased if infraclavicular nerve block is administered, compared to axillary brachial plexus block, for surgical interventions at the level or distal to the elbow.

DETAILED DESCRIPTION:
Pneumatic tourniquets are often used in orthopedic surgery to ensure bloodless surgical field. Besides their obvious positive effects, arterial tourniquets have some unfavorable properties. One of these is tourniquet pain, which can manifest in the presence of an otherwise adequate neuraxial or peripheral nerve block. If it develops, it is usually difficult to manage, and can be severe enough to necessitate conversion to general anaesthesia.

In the past the incidence of tourniquet pain, associated with different nerve blocks has been estimated in clinical trials for which it was a secondary outcome measure. One recent meta-analysis addressed the question: is infraclavicular block (ICB) associated with a lesser incidence of tourniquet pain compared to other brachial plexus blocks. The studies selected by this meta-analysis used different types of nerve block. However it did not address the clinically relevant question: using standard techniques for ultrasound guided brachial plexus block (USgBPB) is the infraclavicular approach associated with a lesser incidence of tourniquet pain than the axillary approach? The following nerves contribute to the perception of tourniquet pain: musculocutaneous, radial, medial cutaneous brachial (MCBN) and intercostobrachial (ICBN). The potential advantage of the ICB over the axillary brachial plexus block (ABPB) in regards to tourniquet pain comes from anatomical reasons. In the pyramid shaped infraclavicular space the cords are much closer to each other; thus the likelihood of achieving effective MCBN and ICBN block is greater. The infraclavicular route has proven to result in an equally effective, reliable and safe block of the brachial plexus, compared to the axillary approach. We hypothesize that the incidence of tourniquet pain is less with infraclavicular block compared to axillary brachial plexus block.

The aim of the study is, to compare the incidence and severity of tourniquet pain associated with ultrasound guided ICB and ABPB in patients undergoing orthopedic surgery at the level or distal to the elbow, with a tourniquet time longer than 45 minutes.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Orthopedic surgery at the level or distal to the elbow
* Expected tourniquet time > 45 min (K-wiring not suitable)

Exclusion Criteria:

* Contraindication of regional anaesthesia, patient is allergic to local anesthetics
* Clinically significant cognitive impairment (Minimental state score < 24)
* Chronic pain syndrome
* Preexisting nerve damage in the operated arm (sensory or motor deficit)
* Axillary clearance in the past
* History of peripheral neuropathy)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-03; Primary Completion 2017-05-09 (Actual); Study Completion 2017-05-09 (Actual)

PRIMARY OUTCOMES:
Incidence of tourniquet pain | Intraoperative period

SECONDARY OUTCOMES:
Onset time of tourniquet pain | Intraoperative period
Severity of tourniquet pain | Intraoperative period
  Mild tourniquet pain (no need for intervention*) Moderate tourniquet pain (need for fentanyl / additional sedation*) Severe tourniquet pain (requiring GA*)
  *: based on the clinical judgement of the responsible clinician (not a member of the study team)
Incidence of adverse events | During block placement
  Vascular puncture or paresthesia during block placement
Block performance time | During block placement
  From commencing sterile preparation to completion of injection of local anaesthetic
Block onset time | 30 minutes after block placement
  From completed injection of local anaesthetic until loss of cold sensation in distribution of radial, ulnar, median and musculocutaneous nerve in the hand and forearm
Incidence of block failure | 30 minutes after block placement
  Presence of cold sensation in at least one distribute of radial, ulnar, median and musculocutaneous nerves in the hand and forearm at 30 min after completion of injection of local anaesthetic

CONTACTS AND LOCATIONS:
Overall Officials: George Shorten, Professor, Study Chair — Professor of Anaesthesia and Intensive Care Medicine, Consultant Anaesthetist, University College Cork / Cork University Hospital; Gabriella Iohom, Dr., Study Director — Consultant Anaesthetist, Senior Lecturer, Cork University Hospital / University College Cork
Locations (1):
- Division of Anaesthesia and Intensive Care, Cork University Hospital, Cork, Co. Cork, Ireland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kam PC, Kavanagh R, Yoong FF. The arterial tourniquet: pathophysiological consequences and anaesthetic implications. Anaesthesia. 2001 Jun;56(6):534-45. doi: 10.1046/j.1365-2044.2001.01982.x. PMID 11412159
- [Background] Estebe JP, Davies JM, Richebe P. The pneumatic tourniquet: mechanical, ischaemia-reperfusion and systemic effects. Eur J Anaesthesiol. 2011 Jun;28(6):404-11. doi: 10.1097/EJA.0b013e328346d5a9. PMID 21502865
- [Background] Sauter AR, Smith HJ, Stubhaug A, Dodgson MS, Klaastad O. Use of magnetic resonance imaging to define the anatomical location closest to all three cords of the infraclavicular brachial plexus. Anesth Analg. 2006 Dec;103(6):1574-6. doi: 10.1213/01.ane.0000242529.96675.fd. PMID 17122242
- [Background] Chin KJ, Alakkad H, Adhikary SD, Singh M. Infraclavicular brachial plexus block for regional anaesthesia of the lower arm. Cochrane Database Syst Rev. 2013 Aug 28;2013(8):CD005487. doi: 10.1002/14651858.CD005487.pub3. PMID 23986434
- [Derived] Brenner D, Iohom G, Mahon P, Shorten G. Efficacy of axillary versus infraclavicular brachial plexus block in preventing tourniquet pain: A randomised trial. Eur J Anaesthesiol. 2019 Jan;36(1):48-54. doi: 10.1097/EJA.0000000000000928. PMID 30461447